CLINICAL TRIAL: NCT00000580
Title: Interruption of Maternal-to-Infant Transmission of Hepatitis B by Means of Hepatitis B Immune Globulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 300; P01HL009011-18A1 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-01

CONDITIONS: Hepatitis B; Hepatitis, Viral, Human; Liver Diseases
MeSH Terms: conditions — Hepatitis B; Hepatitis, Viral, Human; Liver Diseases | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: immunoglobulins, intravenous

SUMMARY:
To evaluate whether hepatitis B immune globulin with a high level of antibody against the hepatitis B antigen would be capable of interrupting maternal-fetal transmission of hepatitis B virus, the single most important route of hepatitis spread in the entire Third World.

DETAILED DESCRIPTION:
BACKGROUND:

A baseline study on the vertical transmission of hepatitis B virus in Taiwan revealed that 15 percent of all pregnant women were persistent carriers of hepatitis B antigen and that 40 percent of their new babies developed a protracted antigenemia during the first 6 months of life. The incidence of acute hepatitis, cirrhosis, and hepatoma was high in Taiwan, and patients with these disorders had a fivefold to sixfold higher prevalence of hepatitis B antigen than healthy persons. Given the important public health problems of this disease in Taiwan and the rest of the Third World, this trial sought to answer the important question of whether hepatitis B immune globulin with a high level of antibody against the antigen would be of utility in combating the problem.

Two hundred and five babies were accepted into the study, which was actually conducted on Taiwan through a contract to the Community Blood Council of Greater New York. Only those babies born of mothers who had HBsAg complement fixation titers of 1:8 or greater were included in these studies. At birth, blood was obtained from the mothers and cord blood from the infants. Follow-up bloods were obtained from both the mother and baby when the infants were 1, 3, 6, 12, 24 and 36 months of age. In addition, all household family contacts were bled at least once during this period.

DESIGN NARRATIVE:

Randomized, double-blind, fixed sample. A total of 205 neonates were assigned to treatment with high-titer hepatitis B immune globulin, standard immune globulin, or albumin placebo within 72 hours of delivery.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Boy and girl infants, birth to 3 years, born to mothers who were hepatitis B surface antigen carriers.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1975-11; Study Completion 1986-06 (Actual)

REFERENCES:
- [Background] Beasley RP, Stevens CE: Vertical Transmission of HBV and Interruption with Globulin, in Vyas GN, Cohen SN, Schmid R (eds.), Viral Hepatitis: A Contemporary Assessment of Etiology, Epidemiology, Pathogenesis and Prevention. Philadelphia, Franklin Institute Press, 1978, 333-345.
- [Background] Stevens CE, Neurath RA, Beasley RP, Szmuness W. HBeAg and anti-HBe detection by radioimmunoassay: correlation with vertical transmission of hepatitis B virus in Taiwan. J Med Virol. 1979;3(3):237-41. doi: 10.1002/jmv.1890030310. PMID 479860